CLINICAL TRIAL: NCT03474653
Title: Latitude-An Observational Study of Patient Choice and the Urethral Bulking Agent, Bulkamid®, Used for the First Line Treatment for Stress Urinary Incontinence and the Impact on a Subsequent Mid Urethral Sling
Brief Title: LATITUDE An Observational Study of Patient Choice and the Urethral Bulking Agent, Bulkamid®
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Manchester University NHS Foundation Trust (Other Government)
Collaborators: Contura (Industry)
Responsible Party: Sponsor
Other Study IDs: V1 15/12/16
Record Dates: First submitted 2018-03-15; First posted 2018-03-22 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Urinary Incontinence; Stress Urinary Incontinence
Keywords: Stress urinary incontinence; Bulking; Bulkamid
MeSH Terms: conditions — Urinary Incontinence; Urinary Incontinence, Stress

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Latitude 1 (Bulking): Women with first line stress incontinence who choose to have Bulkamid as a treatment
- Latitude 2 (Choice): Women with first line stress incontinence who choose to have any treatment including Bulking.

SUMMARY:
Latitude is an observational study exploring how effective Bulkamid ® is as a first line treatment for women with stress urinary incontinence. Women who choose to have Bulkamid as part of their standard clinical care will be asked to complete questionnaires before and after their surgery so that we can assess how their urinary symptoms change.

As a second part of the study, we are asking all patients having any first line treatment for stress incontinence to complete a short questionnaire telling us how they decided what treatment to have. A small number of these women will be contacted via telephone and asked whether they would mind being interviewed to tell us more about this.

We will also interview a number of doctors taking part in Latitude to find out how they counsel patients about different treatment options for stress urinary incontinence.

DETAILED DESCRIPTION:
This is a multi-centre observational study to investigate the effectiveness of the urethral bulking agent, Bulkamid®, as a primary treatment for stress urinary incontinence (SUI). It also contains an embedded qualitative sub-study to investigate factors that influence patient choice of surgical treatment for SUI.

Bulkamid® is a non-toxic hydrogel that is injected under the lining of the urethra. It increases the urethral 'bulk', hence increasing resistance against leakage of urine. It is being increasingly offered as a primary treatment for SUI due to the reduced associated risks, ability to administer in the outpatient setting and recent controversy surrounding polypropylene mesh. However, there is currently limited data on how effective it is as a first line treatment, both in the short and long term, and what effect it may have on secondary continence procedures.

This study aims to collect data from 220 women who choose Bulkamid® as their primary treatment over a total of 60 months to review its effectiveness. Telephone consultations will take place at regular intervals using validated questionnaires to assess SUI symptoms.

It is not known how easy women find it to choose between the surgical treatment options for SUI, what factors they weigh up or what information would help them make this decision. The embedded qualitative study of patient choice will use a combination of questionnaire and 2 in-depth semi structured interviews to investigate this further. Consultant Urogynaecologists will also be interviewed to compare factors they think are important to their patients' treatment decision with what is expressed by women with SUI. The overall aim is to develop a prototype decision aid to better support women when making this treatment decision.

ELIGIBILITY:
Inclusion Criteria:

* All women with urodynamic stress incontinence that are eligible for surgery for SUI.
* Evidence of previous supervised pelvic floor muscle training

Exclusion Criteria:

* OAB (overactive bladder) predominant mixed incontinence
* Any previous surgery for urinary incontinence
* Concomitant prolapse surgery
* Detrusor over activity on urodynamics
* Residual urine > 100ml at urodynamics
* Bladder capacity < 300 ml
* An acute urinary tract infection (UTI)
* An allergic reaction to the local anaesthesia used in the treating unit
* An allergic reaction to all the antibiotics which could be used for prophylaxis
* Current treatment with systemic corticosteroids
* Pregnancy
* Active autoimmune or connective tissue diseases
* Not fluent in English requiring an independent interpreter

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women with urodynamic stress incontinence who wish to proceed with further treatment
Sampling Method: Non-Probability Sample
Enrollment: 399 (Actual)
Dates: Start 2017-06-12 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
PGI-S | 12 months post Bulkamid
  The primary outcome will be the score of PGI-S of patients 12 months after Bulkamid® or the last PGI-S recorded for those who have gone on to have a second injection of Bulkamid® or MUS.

SECONDARY OUTCOMES:
Post Bulking MUS rate | 6, 12, 24 and 60 months
  The number of women who go to have a MUS
Complications post Bulkamid | 6, 12, 24 and 60 months
  Number of women who started taking drugs for OAB after surgery Number of women with recurrent UTI (defined as 2 UTIs in 6 months); Number of women performing clean intermittent self-catheterisation (CISC).
PGI-I; a single question with a 7-item response. | 6, 12, 24 and 60 months
  Patient Global Impressions of Improvement validated questionnaire Number of women with recurrent UTI (defined as 2 UTIs in 6 months); Number of women performing clean intermittent self-catheterisation (CISC).
PGI-S; a single question with a 4-item response. | 6, 12, 24 and 60 months
  Patient Global Impressions of Severity validated questionnaire Number of women with recurrent UTI (defined as 2 UTIs in 6 months); Number of women performing clean intermittent self-catheterisation (CISC).
ICIQ-SF | 6, 12, 24 and 60 months
  International Consultation on Incontinence Questionnaire - Short Form ICIQ-SF; a short 4 question
Electronic Patient Questionnaire | 6, 12, 24 and 60 months
  ePAQ incontinence domains (Pain; Voiding; OAB; SUI; QoL).
Pads used due to leakage | 6, 12, 24 and 60 months
  Number of women still using pads due to leakage question
Pads used due to fear of leakage. | 6, 12, 24 and 60 months
  Number of women still using pads due to fear of leakage question
EQ-5D | 6, 12, 24 and 60 months
  EQ-5D is a standardised measure of health status developed by the EuroQol Group in order to provide a simple, generic measure of health for clinical and economic appraisal

CONTACTS AND LOCATIONS:
Overall Officials: Fiona M Reid, Principal Investigator — Manchester University Hospitals NHS Foundation Trust
Locations (1):
- Manchester University Hospital NHS Foundation Trust, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Data will not be shared with other researchers.